CLINICAL TRIAL: NCT00303667
Title: Reduced Intensity Haploidentical Hematopoietic Stem Cell Transplantation (HSCT) Supplemented With Donor Natural Killer (NK) Cell Infusions in Patients With High Risk Myeloid Malignancies Who Are Unsuitable for Fully Myeloablative Transplantation
Brief Title: Donor Natural Killer Cells and Aldesleukin in Treating Patients w/High Risk AML Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS042; UMN-MT2003-23 (Other: Blood and Marrow Transplantation Program); UMN-IRB-0405M60481 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Acute Myelogenous Leukemia
Keywords: NK cells; natural killer cells; immunotherapy; hematopoietic cell transplant; acute myelogenous leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — aldesleukin; Interleukin-2; IL32 protein, human; Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation; thymoglobulin; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCT w/Donor Natural Killer Cells - short schema (Experimental): Patients with high risk myeloid malignancies undergoing allogeneic hematopoietic stem cell transplantation, receiving fludarabine phosphate (daily dose of 40mg/m^2), cyclophosphamide (administered on Day -15 only), cyclosporin A, total body irradiation, natural killer cells, aldesleukin, and thymoglobulin.
  Interventions: Biological: aldesleukin; Biological: natural killer cells; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total body irradiation; Biological: Thymoglobulin; Drug: Cyclosporin A
- SCT w/Donor Natural Killer Cells - extended schema (Experimental): Patients with high risk myeloid malignancies undergoing allogeneic hematopoietic stem cell transplantation, receiving fludarabine phosphate (daily dose of 35mg/m^2), cyclophosphamide (administered on Days -15 and -16), cyclosporin A, total body irradiation, natural killer cells, aldesleukin, and thymoglobulin.
  Interventions: Biological: aldesleukin; Biological: natural killer cells; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total body irradiation; Biological: Thymoglobulin; Drug: Cyclosporin A; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin — Administered subcutaneously (SQ) 9 million units every other day beginning Day -12 through -2 (evening of natural killer cell infusion) for a total of 6 doses.
  Other Names: Interleukin-2; IL-2
Biological: natural killer cells — Infusion given on Day -12; The targeted infused cell dose of CD3- CD19- selected NK product is within the range of 2-3 x 10^7 cells/kg.
  Other Names: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide — Administered intravenously (IV) 50 mg/kg on Day -15
  Other Names: Cytoxan
  Arms: SCT w/Donor Natural Killer Cells - short schema
Drug: fludarabine phosphate — Administered intravenously (IV) 40 mg/m^2 on Days -18 through -14
  Other Names: Fludara
  Arms: SCT w/Donor Natural Killer Cells - short schema
Procedure: allogeneic hematopoietic stem cell transplantation — On day 0, patients will receive an allogeneic transplant using pool cells from the day -1 and day 0 PBSC which will be CD34+ selected as the donor graft. The graft will be infused over 15-60 minutes.
  Other Names: PBSC
Radiation: total body irradiation — Administered on Day -13, 200 cGy two times.
Biological: Thymoglobulin — intravenous (IV) 3 mg/kg on Day 0 (day of donor CD34 cell infusion)
  Other Names: rabbit ATG
Drug: Cyclosporin A — 1.5 mg/kg by mouth or intravenously for target dose range of 150-250; day -15 through day -8.
  Other Names: CSA
Drug: cyclophosphamide — Administered intravenously (IV) 50 mg/kg on Days -16 and -15
  Other Names: Cytoxan
  Arms: SCT w/Donor Natural Killer Cells - extended schema
Drug: fludarabine phosphate — Administered intravenously (IV) 35 mg/m^2 on Days -18 through -14
  Other Names: Fludara
  Arms: SCT w/Donor Natural Killer Cells - extended schema

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine phosphate and cyclophosphamide, and total body irradiation, before peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer (NK) cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving IL-2 (aldesleukin) after NK cell infusion may stimulate them to kill any remaining cancer cells.

PURPOSE: This phase I/II (currently enrolling in phase II) trial is studying how well a donor natural killer cell infusion works in treating patients who are undergoing donor stem cell transplant for acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the disease-free survival at 6 months and 1 year in patients with high-risk myeloid malignancies who undergo a reduced-intensity haploidentical hematopoietic stem cell transplantation (HSCT) supplemented with donor natural killer (NK) cells.

Secondary

* To evaluate the in vivo expansion of a donor CD3- CD19- selected NK cell product administered after a preparative regimen of cyclophosphamide, fludarabine, and total body irradiation (TBI) and HSCT in these patients.
* To determine the rate of graft failure defined by absolute neutrophil count (ANC) < 500/mm³ by day 28.
* To determine the incidence of grade III-IV acute graft-versus-host disease (GVHD) at 6 months.
* To determine the rate of treatment-related mortality at day 100.
* To determine the incidence of chronic GVHD at 12 months.
* To determine the incidence of disease relapse at 12 months.
* To determine the incidence of post-transplant lymphoproliferative disorder at 12 months.

Correlative

* To correlate immune reconstitution of the in vivo expanded haploidentical NK cells with clinical outcomes.

OUTLINE: This is an open-label study.

Patients receive fludarabine intravenous (IV) over 1 hour on days -18 to -14 and cyclophosphamide IV over 2 hours on days -16 and -15. Patients receive cyclosporin A on Day -15 through Day -8. Patients undergo total body irradiation on day -13. Patients then receive an infusion of donor natural killer cells on day -12 and interleukin-2 subcutaneously on alternating days between days -12 to -2. Patients receive thymoglobulin (ATG) and undergo allogeneic peripheral blood stem cell transplantation on day 0.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* 4.2 High risk acute myeloid leukemia (AML) fitting within one of the following disease groups:

  * Primary induction failure defined as no complete remission (CR) after two or more induction cycles. For primary induction failure (PIF) or refractory AML, the patient must have <5% circulating blasts (and <1000 absolute circulating blasts) beyond Day 28 after last chemo. During work-up period if circulating blasts rise above these levels, the patient is ineligible. The use of hydrea or other non-induction cytotoxic agents is not allowed to reduce blasts and achieve this eligibility. If the blasts are higher than these limits, the patient should be treated on an alternative therapeutic protocol or receive another reinduction attempt. (See section 7 regarding final check of blast status within 7 days of preparative regimen start).
  * Relapsed AML with low disease burden must have less than 5% marrow blasts at time of enrollment for patients who did not receive re-induction or measured at least 28 days from the start of reinduction therapy for patients who did receive re-induction (maximum of 2 re-induction attempts). Patients who have relapsed more than 12 months following a prior HCT and did not reach CR following one re-induction cycle but have less than 10% marrow blasts are eligible.
  * CR3 or greater. This will include CRp defined as CR without platelet recovery to 100,000/mcL.
  * CR1 or CR2 with high risk features (therapy induced, prior myelodysplastic syndrome [MDS] or myeloproliferative disease [MPD], high risk cytogenetic or molecular phenotype) with no available alternate (sibling, unrelated donor [URD] or umbilical cord blood [UCB]) donors.

Patients with prior central nervous system (CNS) involvement are eligible provided that it has been treated and CFS must be clear for at least 2 weeks prior to enrollment.

* Available related HLA-haploidentical donor (3-5 of 6 HLA, A, B and DRB1 matched)
* Karnofsky performance status > 50
* Pulmonary Function: oxygen saturation ≥ on room air and diffusion lung capacity for carbon monoxide (DLCOcor) ≥ 40%
* Cardiac Function: Ejection fraction (EF) ≥ 30%, no uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Able to be off prednisone or other immunosuppressive medications for at least 3 days prior to Day 0
* Women of child bearing potential must have a negative pregnancy test within 14 days prior to study registration and agree to use adequate birth control during study treatment
* Human anti-mouse antibody (HAMA) monitoring: All subjects will be questioned about prior exposure to antibody therapy (including OKT3, rituximab, trastuzumab, etc).

  * For subjects with no prior antibody therapy exposure, no further action will be taken
  * For subjects who have received previous antibody therapies 10 ml of serum will be drawn before starting therapy. The presence of HAMA will not preclude proceeding with treatment.
* Voluntary written consent signed before performance of any study related procedure not part of the normal medical care.

Exclusion Criteria:

* Biphenotypic leukemia
* New or progressive pulmonary infiltrates on screening chest x-ray or chest computed tomography (CT) scan that has not been evaluated with bronchoscopy, if feasible. Infiltrates attributed to infection must be stable/improving (with associated clinical improvement) after 1 week of appropriate therapy (2 weeks for presumed or documented fungal infections). Surgical resection waives any waiting requirements.
* Uncontrolled bacterial or viral infections. Chronic asymptomatic viral hepatitis is allowed.
* Known hypersensitivity to any of the study agents used
* Received other investigational drugs within the 14 days before enrollment

Donor Selection:

* 12-75 years of age
* > 40 kilogram body weight
* In general good health as determined by the evaluating physician
* Donors must be HLA-A, B, DRB1 haploidentical (3-5/6 antigens HLA, A, B, DRB1) match to recipient. Patients and donors will be typed for HLA-A, B and C using at least intermediate resolution DNA techniques for DRB1 at high (allele) resolution. KIR B genotyping will be done on all haploidentical donors, and when feasible, the donor with the most favorable KIR gene profile will be used.
* Able and willing to have up to 4 separate apheresis collections per formed
* Not pregnant
* Human immunodeficiency virus (HIV): HIV-1, HIV-2 negative; HTLV-1, HTLV-2 negative, Hepatitis B and C negative
* Voluntary written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Cooley, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 patients were originally enrolled; only 47 patients were treated. 4 patients received a natural killer cell (NK) infusion but did not get a transplant because of an early death.
Period: Overall Study
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Started | 8 | 39
Completed | 8 | 35 (Completed = remained alive and on study through Day 0 (day of transplant))
Not Completed | 0 | 4
Not completed — Death | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema | Total
Number analyzed (Participants) | 8 | 39 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 36 | 44
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 16 | 20
  Male | 4 | 23 | 27
Region of Enrollment [Number; unit: participants]
  United States | 8 | 39 | 47

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival at 6 Months
Description: Number of patients alive without evidence of disease at 6 months after transplant
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 0 | 4

2. Secondary Outcome: In Vivo Expansion of a Donor NK Cells NK Cell Product
Description: Number of patients with in vivo expansion of donor NK cells. In vivo expansion of NK cell is defined as detection of >100 donor-derived NK cells per microliter of blood.
Time Frame: 12 - 14 days after NK cell infusion
Population: The protocol was amended to add this endpoint after the 8 subjects were enrolled on the short schema. Thus the relevant samples to determine NK expansion were not collected. On the extended schema, 3 of 39 patients died prior to the day on which in vivo donor NK cell expansion was assessed. Thus only 36 patients were evaluable for that endpoint.
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 0 | 36
participants |  | 19

3. Secondary Outcome: Number of Patients With Graft Failure
Description: Number of patients with graft failure defined as <500 donor neutrophils count by day 28 in the absence of residual or relapsed leukemia
Time Frame: Day 28
Population: On the short schema, 1 of the 8 patients, and on the extended schema, 6 of the 39 patients, died prior to Day 28, the day on which engraftment was assessed. Thus, only 7 and 33 patients respectively were evaluable for that endpoint.
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 7 | 33
participants | 1 | 4

4. Secondary Outcome: Incidence of Grade III-IV Acute Graft Versus Host Disease
Description: Grade III-IV acute graft versus host disease is a severe short term complication created by infusion of donor cells into a foreign host
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 0 | 0

5. Secondary Outcome: Number of Patients With Treatment-Related Mortality
Description: Death within the first 100 days related to treatment in patients without relapse or persistent disease.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 1 | 13

6. Secondary Outcome: Incidence of Chronic Graft Versus Host Disease
Description: Chronic graft versus host disease is a severe long term complication created by infusion of donor cells into a foreign host
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 0 | 0

7. Secondary Outcome: Number of Patients With Disease Relapse
Description: Disease relapse is the recurrence of leukemia in patients who had cleared their leukemia after treatment. Patients with persistent leukemia are not evaluable for relapse.
Time Frame: 1 Year
Population: On the extended schema, 16/39 patients either did not clear their leukemia or died before relapse would have been detected (day 28), and thus were not evaluable for relapse.
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 23
participants | 5 | 12

8. Primary Outcome: Disease-free Survival at 1 Year
Description: Number of patients alive without evidence of disease at 1 year after transplant
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 0 | 3

9. Secondary Outcome: Incidence of Post-transplant Lymphoproliferative Disorder (PTLD)
Description: Post-transplant lymphoproliferative disorder (PTLD) is a virally-driven cancer of the lymphoid cells caused by immunosuppressive drugs taken after allogeneic stem cell transplantation to prevent or control graft versus host disease.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | SCT w/Donor Natural Killer Cells - Short Schema | SCT w/Donor Natural Killer Cells - Extended Schema
Number analyzed (Participants) | 8 | 39
participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Up to 3 years post IL-2 infusion.
Description: Adverse event collection for the purposes of this study will focus on targeted adverse events and unexpected adverse events (serious) at specific time points in relation to the NK cell infusion and post NK cell infusion IL-2 injections.
Arm/Group | SCT w/Donor Natural Killer Cells - Extended Schema | SCT w/Donor Natural Killer Cells - Short Schema
Serious Adverse Events (participants affected / at risk) | 38/39 | 8/8
Other Adverse Events (participants affected / at risk) | 39/39 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SCT w/Donor Natural Killer Cells - Extended Schema (N=39) | SCT w/Donor Natural Killer Cells - Short Schema (N=8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 0
Veno-occlusive disease (Hepatobiliary disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Infection with Grade 3 or 4 ANC (Infections and infestations) | 5 | 0
Infection with normal ANC (Infections and infestations) | 6 | 0
Opportunistic infection (Infections and infestations) | 1 | 0
Infection with unknown ANC (Infections and infestations) | 5 | 8
Dysphagia (Gastrointestinal disorders) | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 0
CNS hemorrhage (Nervous system disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Thrombotic microangiopathy (Vascular disorders) | 2 | 0
Other, GI hemorrhage NOS (Gastrointestinal disorders) | 1 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizures (Nervous system disorders) | 0 | 1
Retinal hemorrhage (Eye disorders) | 0 | 1
Demyelinating encephalopathy (Nervous system disorders) | 0 | 1
Neurologic toxicity, NOS (Nervous system disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Fungal infection requiring amputation of a toe (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Neuropathy (Nervous system disorders) | 1 | 0
Altered mental status (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SCT w/Donor Natural Killer Cells - Extended Schema (N=39) | SCT w/Donor Natural Killer Cells - Short Schema (N=8)
Chills (General disorders) | 39 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 4
Edema (General disorders) | 23 | 4
Fatigue (General disorders) | 36 | 6
Fever (General disorders) | 37 | 5
Hypertension (Vascular disorders) | 5 | 0
Hypotension (Vascular disorders) | 7 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Injection Site Reaction (General disorders) | 21 | 0
Myalgia/Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 12 | 6
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 16 | 0
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 18 | 0
Sweats (General disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes